CLINICAL TRIAL: NCT01859780
Title: Visual Distraction as a Means of Enhancing Child Resistance
Acronym: VDCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Laura Bix, Associate Professor, Michigan State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13-246
Record Dates: First submitted 2013-05-01; First posted 2013-05-22 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Unintentional Ingestion of Prescriptions Within Vials and Blisters
Keywords: Poison control; Child resistant packaging; prescription vials; prescription blisters; drug packaging
MeSH Terms: conditions — Blister

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prescription packages (vials and blisters) (Experimental): Stage I Prescription vials and wallets (packaging) with three levels of distractor placement (hidden, absent and obvious) will be tested for an effect of placement on selection behavior and time to package selection.
  Stage II Prescription vials and wallets (packaging) with and without distractors will be tested for an effect on time to open and number of successful openings.
  Interventions: Other: Visual distractor

INTERVENTIONS:
Other: Visual distractor

SUMMARY:
Unintentional poisonings of children continues to be a major issue in the US. According to a study conducted by Cincinnati Children's Hospital Medical Centers, during the period from 2001-2008, emergency room visits for children less than 5 rose 28% as the result of pharmaceutical products. The authors note, "the problem of pediatric medication poisoning is getting worse, not better."

Child resistant closures have been required on most medications sold in the US since the early 1970s. However, most designs attempt to thwart children through purely physical means (e.g. simultaneous dissimilar motion or opening using sequential tasks). Few, if any designs, have utilized perception and cognition as a way to enhance child resistance.

The investigators propose utilizing visual illusions in spaces distinct from the opening mechanism of prescription packages as a means of enhancing child resistance. In this project, visual illusion images are applied to both vials and wallet blisters in order to attract children's interest and prolong the time before opening.

During Stage I, the investigators will determine if the visual distractor attracts attention when samples are displayed in a storage rack. During Stage II, the investigators will test the effect of visual distractors on child resistance as measured by successful openings and time to open.

DETAILED DESCRIPTION:
Stage I

Objective: to determine if the visual distractor attracts attention when samples are displayed in a storage rack.

Eligibility Criteria

To participate in this study children must:

* Be 2 years to 4 ½ years old
* Have parent's permission to be videotaped
* Have parent's signed permission (in the form of the official (IRB approved, signed consent)
* Have no known history of lactose allergy or lactose sensitivity (packages contain a lactose placebo)
* Verbally agree to participate after a brief explanation of what we want them to do

Outcome Measures Categorical variable (package choice) Continuous variable (time to choice)

Stage II Objective: to test the effect of visual distractors on child resistance as measured by successful openings and time to open.

Eligibility Criteria

To participate in this stage of the study children must:

* Have no known history of lactose allergy or lactose sensitivity (packages contain a lactose placebo)
* Be 2 years to 4 ½ years old
* Have their parent's permission to be videotaped
* Have their parent's permission (in the form of the official, IRB approved signed consent)
* Verbally agree to participate after a brief explanation of what we want them to do

Outcome Measures Binary (package opened yes/no) Continuous variable (time to open for those successful)

ELIGIBILITY:
Inclusion Criteria:

* 2-4.5 years of age
* Parental permission to video tape

Exclusion Criteria:

* Lactose allergy or lactose sensitivity

Ages: 2 Years to 54 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 229 (Actual)
Dates: Start 2013-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Package selection | Day of experiment- Stage I
  Selection of one of three treatments in stage one testing (categorical variable)
Time to opening | Day of experiment (Stage II)
  Time it takes a participant to successfully open a given treatment (continuous variable)

SECONDARY OUTCOMES:
Time to selection (continuous variable) | Day of the experiment- Stage I
  Time it takes participants to select package (continuous variable)
Success/Failure to open | Day of the experiment (Stage II)
  Success or failure in opening by package treatment (binary response variable)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Bix, PhD, Principal Investigator — School of Packaging, Michigan State University; Mark Becker, PhD, Principal Investigator — Cognition and Cognitive Neuroscience Group; Judith Danovitch, PhD, Principal Investigator — Knowledge in Development Lab, Psychology
Locations (3):
- United States (3):
  - Packaging Building, East Lansing, Michigan
  - LESA Early Childhood Programs, Howell, Michigan
  - Great Lakes Marketing, Toledo, Ohio

REFERENCES:
- See also: Up and Away Campaign (brochures from this campaign will be sent home with children after testing) — http://www.upandaway.org/